CLINICAL TRIAL: NCT00229944
Title: Randomized, Double-Blind, Controlled Clinical Trial to Compare Efficacy of a Single Dose of Azithromycin Versus a Single Dose of Ciprofloxacin in the Treatment of Adults With Clinically Severe Cholera Due to V. Cholerae O1 or O139
Brief Title: Single Dose Azithromycin in the Treatment of Adult Cholera
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Pfizer (Industry); Tufts Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-022
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-09

CONDITIONS: Cholera
Keywords: Azithromycin; V. cholerae O1 / O139; adults; Bangladesh; Clinical trial
MeSH Terms: conditions — Cholera | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
Cholera remains an important cause of diarrhoeal illness and death in Asia, Africa and Latin America. Antimicrobial therapy is an important adjunct to fluid therapy in the management of patients with cholera, and should be given to all patients with clinically moderate-to-severe disease since they can reduce the diarrhoea duration and stool volume by half. Current therapy for cholera is limited by increasing prevalence of multiply-resistant strains of Vibrio cholerae O1 or O139. Tetracycline and doxycycline had been the drugs of choice for treating cholera, but multiply-resistant strains are now present in all areas where cholera is endemic or epidemic. There is thus a need to identify alternative drugs that are effect in treating this disease.

Azithromycin, a newer macrolide agent, is active in-vitro against V. cholerae, attains high concentrations in the gut lumen, has a long half-life, and is better tolerated than erythromycin, and older macrolide. In this study we will compare efficacy of a single, 1.0 g oral doses of azithromycin and ciprofloxacin in male patients, aged 18-60 years, with cholera due to V. cholerae O1 or O139. Patients with typical "Rice watery" stools of cholera, signs of severe dehydration and characteristic cholera vibrios in a dark-field stool microscopy. Patients who have coexisting illness which may confound assessment of the efficacy or safety will not be eligible. Only those patients who have V. cholerae O1 or O139 isolated from their pre-therapy stool and/or rectal swab culture and remains in the hospital for the entire duration of the study will be eligible for efficacy evaluation. A written informed consent will be obtained from each patients for their enrollment in the study.

Patients will be hospitalized for full 5 days, and asked to return for a follow up evaluation 7 days after discharge. After initial rehydration, patients will be observed for 4 hours, and only those with ³ 20 ml/kg of watery stools during this period will be enrolled for study. Treatment will be random, and blinded to study staff and patients. Clinical success of therapy will be defined as resolution of watery stool within 48 hours of administration of the study drug, and bacteriologic success will be defined as the inability to isolate V. cholerae O1 or O139 from fecal/rectal swab cultures of patients after 48 hours of therapy, i.e. on day 3 and on all subsequent days of the study. Patients in whom therapy clinically fails will be treated for 3 days with an effective alternate drug without opening the study code. Ninety one evaluable patients will be required in each group to show with a power of 80% and a type I error of 5% that the two treatment regimens are equivalent (i.e. the 95% confidence interval for the difference in efficacy between the two groups is not greater than 10%).

If single-dose azithromycin therapy is found effective it will provide an important option for the treatment V. cholerae infections, especially those caused by multiply-resistant strains.

DETAILED DESCRIPTION:
A total of 182 evaluable patients (those with a positive stool culture for V. cholerae O1 or V. cholerae O139 and remain in the study for full 5 days) will be required for this study.

Patients who meet the initial entry criteria will be admitted into the study ward of the ICDDR,B, weighed (Dehydration Weight), assessed for hydration status and rehydrated using an intravenous polyelectrolyte solution ("Dhaka Solution" containing 133 mmol/l of sodium, 13 mmol/l of potassium, 98 mmol/l of chloride and 48 mmol/l of bicarbonate) over a 3-hour period in accordance with the WHO guidelines [53], and re-weighed (Rehydration Weight). Rice-based oral rehydration salts (ORS) solution (sodium 90 mmol/l, potassium 20 mmol/l, chloride 80 mmol/l, bicarbonate 30 mmol/l, and rice powder 50 gram per litre) will be used as the primary maintenance fluid once initial rehydration is accomplished, however, intravenous polyelectrolyte solution will be used as the maintenance fluid for patients with excessive vomiting (usually > 4 episodes per hour) or with rapid stool losses (usually >10 ml/kg.hour), or those who are unable to drink enough ORS solution for maintenance of their hydration. Patients will be allowed to drink plain water ad libitum after the initial rehydration. All fluid intake and output during rehydration (and throughout the study) will be recorded. A stool specimen will be collected from the patients for dark-field microscopic examination to document the presence of V. cholerae.

Following rehydration, stool output will be measured for a 4-hour period in the maintenance phase, to be called "Observation Period", and those with a stool output of ³ 20 ml/kg during this period and those who also have V. cholerae demonstrated in their stool dark-field examination will be considered eligible for enrollment into the study if they provide voluntary informed consent. This observation period will help establish that patients enrolled in the study have moderate to severe disease, so that the potential impact of therapy can be evaluated (as any therapy is likely to appear effective in mild disease).

On final enrollment into the study, a more complete history and physical examination will be performed, and all findings will be recorded on pre-designed data collection forms.

Patients entered into study will be randomly assigned to receive either a single, 1 gram oral dose of azithromycin or a single, 1 gram oral dose of ciprofloxacin. Patients entered into study will be assigned a consecutive study number which will have been previously randomly assigned to one of the two treatment regimens, and this randomization will be done using a computer generated random number list with a fixed block length of 4. Study drugs will be administered after completion of the four-hour observation period, and at least 2 hours after the last food intake. The time of administering study drug will be considered as the beginning (the "0" hour) of the study. For patients who vomit within 10 minutes of ingestion of study drug, the dose of the study drug will be repeated. For this purpose, all study drugs will be available in duplicate. Such events will be recorded, and data of these patients will be carefully evaluated. The study drugs will be prepared in identical form to allow for blinding of treatment. Randomization will be done by Pfizer, USA who will also provide coded study drugs.

Patients will be hospitalized for 5 complete days to be counted from the time of administration of the study drug (Each consecutive, 24-period constituting a day). The following clinical and laboratory evaluations will be done for each of the study patients:

* Body Weight: On initial entry into the study, after initial rehydration, at "0" hour of the study (which will coincide with administration of the study drug), and at 24 hour intervals beginning from the time of administration of study drug.
* History and physical examination: On admission, after initial rehydration, at "0" hour of the study, and at least once daily during hospitalization. This will also include evaluation for potential adverse events.
* Vital signs: Oral temperature, pulse and respiratory rates, and blood pressures will be recorded on admission (dehydrated), after rehydration, at the end of the 4-hour observation period ("0" hour of the study), and every 6 hours after administration of the study drug.
* Measurement of stool volume: Will be done for the rehydration period, the four hour observation period, and for each 6-hour period after administration of study drug.
* Characterization of stool: Individual stool will be categorized as either watery or soft or formed; the worst stool character of each 6 hour study period will be used to categorize that time period.
* Stool culture for V. cholerae O1, O139 and non-Ol; and Shigella and Salmonella: Will be done on admission, on study day two and at follow up.
* Rectal swab culture for V. cholerae O1 and O139: Will be done on admission, and on each study day.
* Hematological studies: Serum electrolytes, creatinine and serum Sp. gr., and haematocrit will be determined before and after rehydration, and 24 hours after administration of the study drug (3.0 ml of blood will be required for these tests each time, i.e. a total of 9.0 ml of blood). Complete blood count, and platelet count will be done just before administration of the study drug, however, this may also be done subsequently only if clinically indicated.
* Pharmacokinetic studies: For the first 40 patients enrolled into the study, venous blood will be obtained for determination of the serum concentration of the study drugs at either of the following time intervals from administration of the study drug- 3, 12, 24 or 48 hours. An indwelling catheter with two way stop cock will be introduced to avoid repeated venipuncture which will be taken off 3 hours after administration of the study drug; all subsequent blood samplings will be done by individual venipunctures. This will require only 1.0 ml of venous blood, and serum will be separated and stored at -70EC until assayed. For determination of stool concentration of the study drugs, aliquots of stool (About 5.0 ml each) will be obtained from stool collected over each 6 hour period during the first two days of the study, and like serum, will be stored and analyzed.
* Handling of Treatment Failures: If the study treatment is judged to have failed clinically patients will be treated for 3 days with an agent other than azithromycin or ciprofloxacin to which the isolate of V. cholerae will be found to be susceptible to. The treatment code will not be broken for these patients. Patients with microbiological failure will be treated with a suitable drug as determined by antimicrobial susceptibility of such isolates.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 60 years
* Gender: Male (To facilitate accurate measurement of stool and urine, and also due to the difficulties in hospitalizing women for longer duration)
* Duration of illness: 24 hours or less
* Written informed consent for participation in the study
* Dehydration status: Signs of severe dehydration as determined by World Health Organization criteria.
* Positive stool dark-field microscopic examination for V. cholerae, and subsequent isolation of V. cholerae O1 or O139 from an admission culture of a stool or rectal swab sample.

Exclusion Criteria:

* History of receiving even one dose of an antimicrobial agent effective in the treatment of cholera, and even a single fose of the drugs under evaluation.
* Concomitant infection requiring antimicrobial therapy other than the study drugs which may interfere with evaluation of either the efficacy or safety of the study drugs.
* A concomitant illness which may confound evaluation of outcome or is a contraindication for use of either of the study drugs (chronic heart, lung, of kidney disease, or instance), or conditions which may confound evaluation of adverse events of the study drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220
Dates: Start 2002-12; Study Completion 2004-05

PRIMARY OUTCOMES:
Clinical success
Bacteriological Success

SECONDARY OUTCOMES:
Rates of clinical and bacteriologic relapse.
Duration of diarrhoea in hours, and duration of fecal excretion of V. cholerae O1 or O139 in days.
Volume of watery/liquid stool for each 6 and 24 hour of the study, and also the total amount of watery/liquid stools during the study period.
Frequency of vomiting and the amount of vomitus, and proportion of patients with vomiting on each study day.
Intake of oral and intravenous fluids for each 24 hour as well as the entire duration of the study.
Proportion of patients with resolution of diarrhoea on each study day.
Proportion of patients with a positive culture for infecting V. cholerae O1 or O139 on each study day.

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Saha, MBBS,MS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Result] Saha D, Karim MM, Khan WA, Ahmed S, Salam MA, Bennish ML. Single-dose azithromycin for the treatment of cholera in adults. N Engl J Med. 2006 Jun 8;354(23):2452-62. doi: 10.1056/NEJMoa054493. PMID 16760445